CLINICAL TRIAL: NCT01084421
Title: A Computer-Based Parent/Adolescent HIV Communication Intervention for Latinos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Antonia M. Villarruel, Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HUM00020148; R21NR010457 (NIH)
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: HIV/AIDS; STD; Pregnancy
Keywords: Adolescents; Parents; Computer Based; Latino; Sexual Communication
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer based intervention (Experimental): Participants receive content about adolescent sexual risk and HIV prevention, strategies to support sexual specific communication and parent-adolescent communication in general.
  Interventions: Behavioral: Computer-based parent-adolescent HIV communication
- Wait list control group (No Intervention): Participants will receive the computer based intervention at 3 months follow-up

INTERVENTIONS:
Behavioral: Computer-based parent-adolescent HIV communication — The parental intervention consists of a 60 minute computer-based program delivered in two sessions (one per week). The DVD ROM provides information about adolescent sexual risk and HIV prevention, strategies to support sexual specific communication and parent-adolescent communication in general. The computer based education program is provided in Spanish.
  Other Names: Cuidalos
  Arms: Computer based intervention

SUMMARY:
The purpose of this study is to examine the efficacy of a brief culturally appropriate and theory-based parental communication intervention designed to improve parent-adolescent sexual communication and reduce adolescent sexual risk behavior.

DETAILED DESCRIPTION:
Latino adolescents are at high risk for contracting HIV/AIDS. Few individual and even fewer parent interventions have been developed to address this persistent problem. Parent communication interventions provide an opportunity to enhance individual adolescent based approaches. However, there is a need for theory and culture based interventions focused on Latino parents. The program implemented in this study was designed for parents, to indirectly help reduce the health risks of their adolescents, including unintended pregnancy and STDs, including HIV/AIDS. The study has three aims regarding the examination of whether the computer based parental communication intervention is 1) associated with a greater increase in parents' comfort with, and quantity of communication; 2) associated with a greater increase in adolescents' intentions to abstain from sex and/or avoid unprotected intercourse and decreased self-reported intercourse and unprotected intercourse; and 3) feasible and acceptable to Spanish dominant Latino parents and their adolescent children.

ELIGIBILITY:
Inclusion Criteria:

* Latino parents who have adolescents 14 to 17 years of age
* Spanish dominant or bilingual

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
general parent-adolescent communication, parent-adolescent sexual risk communication, comfort with communication | pretest, 1 week, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonia M Villarruel, PhD,RN,FAAN, Principal Investigator — University of Michigan
Locations (1):
- Detroit Hispanic Development Corporation (DHDC), Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No